CLINICAL TRIAL: NCT02864095
Title: The Effects of Low-dose Epinephrine Plus Tranexamic Acid on Perioperative Haemostasis and Inflammatory Reaction in Major Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Liu Yang, Professor, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Hip blood
Record Dates: First submitted 2016-07-28; First posted 2016-08-11 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Blood Loss
Keywords: Arthroplasty, Replacement, Hip; Epinephrine; Tranexamic acid
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravenous epinephrine (Experimental): Intravenous (IV) low dose epinephrine
  Interventions: Drug: Tranexamic acid (TXA); Drug: Epinephrine
- Topical epinephrine (Experimental): Topical epinephrine
  Interventions: Drug: Tranexamic acid (TXA); Drug: Epinephrine
- Control (Active Comparator): No epinephrine
  Interventions: Drug: Tranexamic acid (TXA)

INTERVENTIONS:
Drug: Tranexamic acid (TXA) — IV and topical administration
Drug: Epinephrine
  Arms: Intravenous epinephrine; Topical epinephrine

SUMMARY:
The purpose of this study is to compare the blood loss of intravenous and topical administration of low dose epinephrine plus combined administration of intravenous and topical tranexamic acid for primary total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 20 and 75 who were diagnosed with as having osteoarthritis or osteonecrosis of the femoral head
* Scheduled for an elective primary total hip arthroplasty
* Those who were willing and able to return for follow-up over at least a 6-month postoperative period

Exclusion Criteria:

* Acute coronary syndrome < 6 months
* Glaucoma,pheochromocytoma, thyrotoxicosis, digoxin intoxication, serum potassium < 3.0 mmol, alcohol abuse, premenopausal women
* Current treatment with adenosine diphosphate (ADP) receptor antagonists, Factor Xa or thrombin inhibitors,heparin (excluding Low Molecular Weight Heparin (LMWH) for perioperative thromboprophylaxis), tricyclic antidepressants, or monoamine oxidase（MAO) or Catechol-O-methyltransferase (COMT) inhibitors
* Patients with history of thromboembolic disease, bleeding disorder
* Patients with history of renal impairment, cardiovascular diseases (previous myocardial infarction, atrial fibrillation ) or cerebrovascular conditions (previous stroke or peripheral vascular surgery)
* Allergy to TXA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Blood loss on post-operative day 1 | 1 day

SECONDARY OUTCOMES:
Length of hospital stay | 1 months
Number of patients with infection | 1 months
Number of deep vein thrombosis cases | 1 months
Number of pulmonary embolism cases | 1 months
Number of plexus venosus leg muscle thrombosis | 1 months
Serum levels of IL-10（Preoperation, intraoperation and post-operation） | Preoperation, intraoperation and up to 2 days post-operation
Serum levels of IL-6（Preoperation, intraoperation and post-operation） | Preoperation, intraoperation and up to 2 days post-operation
Serum levels of IL-1β（Preoperation, intraoperation and post-operation） | Preoperation, intraoperation and up to 2 days post-operation
Serum levels of TNF-α（Preoperation, intraoperation and post-operation） | Preoperation, intraoperation and up to 2 days post-operation
Haemoglobin (Hb) | 7 days
Hematocrit (Hct) | 7 days
Platelets (PLT) | 7 days
Blood loss on post-operative day 3 | 3 days
Preoperation, intraoperation and post-operation R value (min) of thrombelastogram | Preoperation, intraoperation and up to 2 days post-operation
Preoperation, intraoperation and post-operation K value (min) of thrombelastogram | Preoperation, intraoperation and up to 2 days post-operation
Preoperation, intraoperation and post-operation Angle (deg) of thrombelastogram | Preoperation, intraoperation and up to 2 days post-operation
Preoperation, intraoperation and post-operation MA (mm) of thrombelastogram | Preoperation, intraoperation and up to 2 days post-operation
Preoperation, intraoperation and post-operation comprehensive index of blood clotting (CI) of thrombelastogram | Preoperation, intraoperation and up to 2 days post-operation
Preoperation, intraoperation and post-operation LY30 (%) of thrombelastogram | Preoperation, intraoperation and up to 2 days post-operation
Number of patients with blood transfusion | 7 days
  Number of transfusion cases, number of units transfused and amount of transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided